CLINICAL TRIAL: NCT06387797
Title: Primary and Secondary Prevention of Type 2 Diabetes Mellitus in At-risk and Underrepresented Minority Populations in Clark County Through Enhanced Nutrition Cooking Education
Brief Title: Primary and Secondary Prevention of Type 2 Diabetes Mellitus in Clark County
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: University of Nevada, Reno (Other)
Responsible Party: Principal Investigator, Sara K Rosenkranz, Associate Professor in Kinesiology and Nutrition Sciences, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UNLV-2023-321
Record Dates: First submitted 2024-04-16; First posted 2024-04-29 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: At Risk for Type 2 Diabetes Mellitus; Pre Diabetes
Keywords: pre-diabetes; primary prevention; adults
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two parallel study arms.
  1. Cooking Matters for Adults (CMA) Curriculum Delivery over 6 weeks
  2. CMA + Enhanced cooking classes with added components comprising cooking practices specific to diabetes prevention, online information as well as short assignments and activities regarding sleep, stress, physical activity, and sedentary behaviors. The CMA+ arm will also have the opportunity to use a continuous glucose monitor (CGM) for 10 days immediately following the baseline assessment visit. This will be an optional component and participants will not be excluded if they do not wish to use the CGM. (6 weeks)
Who Masked: Outcomes Assessor
Masking Description: Because of the parallel arm differences, it would not be possible to mask the arm assignment for the participant or investigator. However, we will mask the arm assignment for the outcomes assessor, in particular for the HbA1c% assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cooking Matters for Adults (CMA) (Active Comparator): Arm 1) CMA: 6 didactic sessions delivered once per week for 6 weeks at the UNLV Nutrition Center (in person) Baseline and post-test assessments and 6 cooking classes.
  * Lesson 1: Let's Get Cooking!
  * Lesson 2: Choosing Fruits, Vegetables and Whole Grains
  * Lesson 3: Healthy Starts at Home
  * Lesson 4: The Power of Planning
  * Lesson 5: Shopping Smart
  * Lesson 6: Recipes for Success
  Interventions: Behavioral: Cooking Matters for Adults (CMA)
- Cooking Matters for Adults (CMA+) (Experimental): Baseline and Post-test assessments and The CMA curriculum + Enhanced cooking classes with added components comprising cooking practices specific to diabetes prevention, online information as well as short assignments and activities regarding sleep, stress, physical activity, and sedentary behaviors. The CMA+ arm will also have the opportunity to use a continuous glucose monitor (CGM) for 10 days immediately following the baseline assessment visit. This will be an optional component and participants will not be excluded if they do not wish to use the CGM.
  Interventions: Behavioral: Cooking Matters for Adults (CMA+)

INTERVENTIONS:
Behavioral: Cooking Matters for Adults (CMA+) — Six cooking classes + enhanced elements, such as diabetes-specific nutrition and cooking information, and online educational information as well as short assignments and activities regarding sleep, stress, physical activity, and sedentary behaviors. This arm will have the opportunity to use a continuous glucose monitor (CGM) for 10 days immediately following the baseline assessment. Each week, participants will collect their own fecal samples in the privacy of their own homes and will return them at their next cooking class. They will also complete a final fecal sample before the follow-up. Finally, 6-weeks after completion of the cooking classes, researchers will follow up via phone, email, or Zoom (participants will provide their preferred method of contact) to complete follow-up assessments of current lifestyle practices and barriers to fruit and vegetable consumption.
  Arms: Cooking Matters for Adults (CMA+)
Behavioral: Cooking Matters for Adults (CMA) — Participants will attend cooking and educational sessions once per week for 6 weeks. In addition, they will receive recipes and produce boxes with instructions to prepare the recipe at some point prior to their next class. They will also be invited to the online Google Classroom site where all intervention materials will be housed for their convenience. Each week, participants will collect their own fecal samples in the privacy of their own homes and will return them at their next cooking class. They will also complete a final fecal sample before the follow-up (kits provided at the final cooking class, for a total of 6 fecal samples per participant). Finally, 6-weeks after completion of the cooking classes, researchers will follow up via phone, email, or Zoom (participants will provide their preferred method of contact) to complete follow-up assessments of current lifestyle practices and barriers to fruit and vegetable consumption.
  Arms: Cooking Matters for Adults (CMA)

SUMMARY:
This pilot and feasibility study aims to assess the effectiveness of a nutrition education intervention using the Cooking Matters for Adults Curriculum (SNAP-Ed). The study compares this standard curriculum with an enhanced version that includes the same curriculum but has additional components, incorporating specific information related to type 2 diabetes. Additionally, participants in the enhanced group will receive continuous glucose monitors to wear during the study for 10 days. The primary outcomes of the study include evaluating the acceptability of the intervention, and the feasibility of conducting the intervention at the UNLV Nutrition Center. The investigators will also assess participants' Knowledge, Attitudes, and Intentions regarding produce consumption. Alongside feasibility and acceptability, the study aims to explore the preliminary effectiveness of the intervention in increasing fruit and vegetable consumption, reducing HbA1c, managing cardiometabolic risk, and improving gut microbiome composition and diversity among participants in the program. The investigators will also assess changes in other lifestyle behaviors from baseline to post-intervention (6 weeks) (sleep, stress, physical activity, and sedentary behavior).

DETAILED DESCRIPTION:
The long-term goal of this study is to reduce the healthcare costs and burdens associated with T2DM among at-risk populations in Nevada by reducing the incidence of type 2 diabetes mellitus. For the current study, the investigators will determine the feasibility and acceptability of this 6-week intervention. Short-term objectives for the current pilot and feasibility study include developing recruitment, screening, and delivery processes through UNLV's Nutrition Center to improve future extramural grant applications. The investigators hope to have preliminary data regarding whether or not a 6-week enhanced diabetes prevention nutrition education intervention (with education about multiple lifestyle behaviors) is more effective than the basic CMA curriculum for improving cardiometabolic health outcomes that represent risk for developing type 2 diabetes. Additionally, the investigators are using feedback tools to help participants in the enhanced study arm to see their continuous glucose levels in real-time, and to understand the composition of their gut microbiome via collection of stool swab samples.

Baseline Assessments will include:

Finger-sticks for lipids, glucose, and HbA1c%, BIA body composition assessments including height and weight, waist circumference, blood pressure, and questionnaire completion.

Questionnaires will include:

Health History Questionnaire Physical activity and sedentary behavior (IPAQ-short form) (10-15minutes) Dietary intake (3-day dietary recall via ASA24) (Online-15 minutes for each recall) Stress (PSS-10) (10minutes) Sleep quantity and quality (Pittsburgh Sleep Quality Index and Sleep Hygiene Index) (10-15 minutes) Nutrition security screener (5minutes) In addition to these questionnaires, participants will be asked to complete standard questions that are used in the CMA curriculum.

An accelerometer will be secured via an adhesive pocket attached to the front upper thigh, for at least 7 days from the time participants get up to the time they go to bed.

Following baseline assessments, participants will be randomized to the CMA only or the CMA+ arm of the study. Participants randomized to the CMA+ arm will also have a CGM attached to their upper arm (non-dominant hand). Once at least 20 participants have been enrolled, the cooking classes will be scheduled in cohorts of 12-15 participants per study arm, based on limited capacity in the Nutrition Center kitchen. Multiple cohorts will be enrolled during the 2-year period of the grant up to enrollment of 120 participants.

The CMA Curriculum will be used for both arms of the intervention. Participants will attend cooking and educational sessions once per week for 6 weeks. In addition, participants will receive recipes and produce boxes with instructions to prepare the recipe at some point prior to their next class. Participants will also be invited to the online Google Classroom site where all intervention materials (according to the study arm they are randomized to) will be housed for their convenience. Each week, participants will collect their fecal samples in the privacy of their own homes and will return them at their next cooking class. Investigators will provide paper bags that are opaque for privacy for participants to use for returning their samples. Participants will also complete a final fecal sample before the follow-up (kits provided at the final cooking class, for a total of 6 fecal samples per participant in the CMA+ arm). Using a basic collection scoop in a DNA/RNA shield is recommended for this purpose.

The CMA+ arm will also use the CMA Curriculum, but will also include enhanced elements, such as diabetes-specific nutrition and cooking information, and online educational information as well as short assignments and activities regarding sleep, stress, physical activity, and sedentary behaviors. The CMA+ arm will also have the opportunity to use a continuous glucose monitor (CGM) for 10 days immediately following the baseline assessment visit. This will be an optional component and participants will not be excluded if they do not wish to use the CGM.

For both arms, the Google Classrooms platform will be used to house curriculum materials, allow for social interaction and questions to the researchers, and will include videos of cooking demonstrations, ideas for the enhanced arm about how to implement strategies for behavior change for lifestyle behaviors (sleep, physical activity, dietary intake, sedentary behavior, and stress).

Follow-up (at 6 weeks):

Following the completion of the 6-week intervention period, follow-up assessments will be conducted again via appointment at BHS 343 (these will be identical to the baseline assessment visit without the CGM or informed consent processes. Additionally, only 1 24-hour food recall will be conducted at this follow-up visit. These procedures will include Finger-sticks for lipids, glucose, and HbA1c%, BIA body composition assessments including height and weight, waist circumference, blood pressure, and questionnaire completion. Finally, 6-weeks after completion of the cooking classes, researchers will follow up via phone, email, or Zoom (participants will provide their preferred method of contact) to complete follow-up assessments of current lifestyle practices and barriers to fruit and vegetable consumption. This will allow investigators to determine preliminary adherence to any changes from baseline.

If a participant discontinues their participation in the study, any data collected up to that point will be retained for analysis, following the intent-to-treat principle. Since blood will only be collected through finger-stick samples, these will be immediately analyzed upon collection, and the blood will be safely disposed of in a biohazard container. Sharps will be discarded in designated sharps containers. There will be no storage of plasma or blood samples.

All data will be promptly entered into the study database and will be identified solely by a unique study ID number (a randomly generated 3-digit code combined with the study abbreviation and visit number). To ensure confidentiality, all data will be deidentified for storage (electronic and paper-based) public presentations and subsequent publications. Any personally identifiable information will be stored exclusively in hard copy, within a locked file cabinet, accessible only to the Principal Investigator and authorized study personnel. The CMA comprises 6 nutrition education workshops. Over the 2-year study period. We will deliver a series of 5 sessions (2 months duration) including 2 cohorts in each session, for a total of 10 cohorts of 12-15 participants. The sessions will be led by a Nutrition Sciences graduate student who is seeking the Registered Dietitian Nutritionist (RDN) credential or who already holds the RDN credential.

Arm 1) CMA: 6 didactic sessions delivered once per week for 6 weeks

* Lesson 1: Let's Get Cooking!
* Lesson 2: Choosing Fruits, Vegetables and Whole Grains
* Lesson 3: Healthy Starts at Home
* Lesson 4: The Power of Planning
* Lesson 5: Shopping Smart
* Lesson 6: Recipes for Success

Arm 2) CMA+: 6 didactic sessions + Enhanced cooking classes with added components comprising cooking practices specific to diabetes prevention, strategies for increasing self-efficacy for fruit and vegetable consumption, and weekly produce distribution.

o After completion of the program, participants who are eligible will be referred to a DSMPE, diabetes nutrition education and cooking classes (6 weeks) through the Southern Nevada Health District.

• Six weeks after intervention completion, we will follow-up with program participants through phone and/or email to determine sustainability of any behavioral changes, and to better understand barriers to fruit and vegetable consumption.

ELIGIBILITY:
Inclusion Criteria:

People with pre-diabetes, or those self-identifying as at-risk for type 2 diabetes mellitus (T2DM).

Risk for T2DM can be determined through indicators such as family history of T2DM, overweight or obesity, metabolic syndrome, HbA1c levels between 5.7% and 6.4%, or fasting blood glucose levels between 100 and 125 mg/dL. There is increased risk for T2DM among American Indian/Alaska Native, Black and Hispanic adults as compared with White and Asian adults; adults ages 25 and older with less than a high school education, as compared with those with higher education levels; and adults ages 25 and older with household incomes less than $25,000 as compared with those with higher income levels.

Exclusion Criteria:

People who have been diagnosed with T2DM or tested at an HbA1c% level that indicates T2DM. (>6.4%) People who are non-English speaking (this is a feasibility/pilot study, if effective we will propose a fully-powered trial that we plan to translate into Spanish). The curriculum we are using has a Spanish version that we can make available if needed once a participant is enrolled. Additionally, the study coordinator is a student listed on this application who is fluent in Spanish and can help those with limited English capability to ensure participants understand the study and what is expected.

People who are unable to attend in-person cooking classes at the UNLV Nutrition Center for 6 weeks using their own means of transportation.

People who are unwilling to undergo multiple finger-sticks for determining HbA1c, lipids, and glucose levels.

Anyone who has been diagnosed with cardiovascular or metabolic diseases, and or using medications currently to control blood glucose, including Metformin or insulin.

People who have uncontrolled high blood pressure (SBP: >=140/DBP >=90) People who have implantable metal; (e.g., pacemaker) because body composition will be measured via bioimpedance.

People who are actively trying to lose weight, or currently enrolled in a weight loss program or other dietary intervention.

People who have dietary restrictions including those following a vegan diet, gluten-free diet, or with food allergies to any fruits or vegetables.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of conducting the intervention | At one year
  Study team will analyze rate and success with recruiting, retention in the study, completion, adherence to protocol
Acceptability of the intervention | At 6-weeks
  Participant will rate the intervention overall for acceptability
Acceptability of each cooking class | week 1, week 2, week 3, week 4, week 5, and week 6
  Participants will rate each cooking class for acceptability

SECONDARY OUTCOMES:
Knowledge about the importance of produce consumption | baseline and week 6
  questionnaire that asks about understanding of the produce consumption for preventing diabetes
Attitudes toward produce consumption | baseline and week 6
  questionnaire asking about positive or negative perceptions of produce consumption for prevention of diabetes
Intentions to consume recommended amounts of produce during and after intervention | baseline and week 6
  questionnaire that asks for ratings of intention to consume recommended amounts of produce
Changes in fruit and vegetable consumption in servings per day | baseline and week 6
  questionnaire of servings of fruits and vegetables consumed per week
HbA1c% | baseline and week 6
  hemoglobin A1c% from fingerstick
Body weight in kg | baseline and week 6
  body weight measured using SECA bio-electrical impedance scale
Gut Microbiota composition | week 1, week 2, week 3, week 4, week 5, and week 6
  ratio of beneficial/harmful bacteria and microbiota alpha and beta-diversity from participant stool samples
waist circumference in cm | baseline and week 6
  waist circumference measured via tape measure
body fat percentage (%) | baseline and week 6
  body fat percentage determined via SECA bio-electrical impedance scale
non fat mass in kg | baseline and week 6
  amount of mass that is not body fat determined by SECA bio-electrical impedance scale

OTHER OUTCOMES:
blood pressure in mmHg | baseline and week 6
  blood pressure assessment via automated blood pressure device
fasting blood glucose in mg/dL | baseline and week 6
  fasting blood glucose via capillary whole blood from a fingerstick
fasting total cholesterol in mg/dL | baseline and week 6
  fasting total cholesterol via capillary whole blood from a fingerstick
fasting LDL cholesterol in mg/dL | baseline and week 6
  fasting LDL cholesterol via capillary whole blood from a fingerstick
fasting HDL cholesterol in mg/dL | baseline and week 6
  fasting HDL cholesterol via capillary whole blood from a fingerstick
fasting triglyceride level in mg/dL | baseline and week 6
  fasting triglyceride level via capillary whole blood from a fingerstick
Usual dietary quality | baseline and post-test
  3-day food recall at baseline via researcher led online ASA24 to determine usual dietary quality, scored via the Healthy Eating Index
Week 6 dietary quality | week 6
  1-day food recall via researcher led online ASA24 to determine dietary quality scored via the Healthy Eating Index
physical activity energy expenditure average kcals per day | baseline and week 6
  Fibion accelerometer attached to upper thigh to measure physical activity energy expenditure
Time spent in sedentary behavior in minutes per day | baseline and week 6
  Fibion accelerometer attached to upper thigh to measure time spent in sedentary behavior and International Physical Activity Questionnaire-Short form (IPAQ-SF)
physical activity intensity distribution as minutes per day and average percentage of day | baseline and week 6
  Fibion accelerometer attached to upper thigh and International Physical Activity Questionnaire-Short form (IPAQ-SF) to measure percentage time spent in different physical activity intensities (light, moderate, and vigorous physical activity)
sleep quantity in hours per day | baseline and week 6
  hours of sleep reported via Fibion accelerometer attached at the front of the thigh and self-report using the Pittsburgh Sleep Quality Index Questionnaire
sleep quality | baseline and week 6
  hours of sleep and quality of sleep reported via accelerometer and self-report using the Pittsburgh Sleep Quality Index Questionnaire and the Sleep Hygiene Index Questionnaire
stress levels | baseline and week 6
  Perceived Stress Scale 10 (PSS-10) questionnaire used to assess stress levels
Nutrition Security | baseline and week 6
  Nutrition security measured via self-report Nutrition Security-Screener questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sara K Rosenkranz, PhD, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- University of Nevada, Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable participant data will be made available to other researchers upon appropriate request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 6 months after publication of the primary outcomes manuscript for a minimum of three years.
Access Criteria: Upon reasonable request to the study PI